CLINICAL TRIAL: NCT06818266
Title: Efficacy and Safety of Tocilizumab for Acute Chest Syndrome Treatment in Pediatric and Adult Patients With Sickle Cell Disease
Brief Title: Efficacy and Safety of Tocilizumab for Acute Chest Syndrome Treatment in Patients With Sickle Cell Disease
Acronym: TOCIACS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220797; 2023-505109-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-09; First posted 2025-02-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
Keywords: Sickle cell disease; Acute chest syndrome; Tocilizumab
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arms A : Tocilizumab (RoActemra®, 20 mg/mL) (Experimental): One single intravenous infusion at 8 mg/kg (up to a maximum of 800 mg) for patients ≥ 30 kg and 12 mg/kg for patients < 30 kg.
  Interventions: Drug: Tocilizumab (RoActemra®, 20 mg/mL).
- Arm B : Placebo (NaCl 0.9%) (Placebo Comparator): One single intravenous infusion
  Interventions: Drug: Placebo (NaCl 0.9%)

INTERVENTIONS:
Drug: Tocilizumab (RoActemra®, 20 mg/mL). — One single intravenous infusion at 8 mg/kg (up to a maximum of 800 mg) for patients ≥ 30 kg and 12 mg/kg for patients < 30 kg
  Arms: Arms A : Tocilizumab (RoActemra®, 20 mg/mL)
Drug: Placebo (NaCl 0.9%) — One single intravenous infusion
  Arms: Arm B : Placebo (NaCl 0.9%)

SUMMARY:
The purpose of this study is to determine whether a single infusion of tocilizumab is effective in reducing the time to successful weaning from both supplemental oxygen and any respiratory support, in pediatric and adult patients with sickle cell disease (SCD) during acute chest syndrome (ACS).

DETAILED DESCRIPTION:
SCD is a severe hemoglobinopathy, considered the first monogenic disease in the world. ACS, one of the most frequent and serious complications of SCD, is the first cause of hospitalization and mortality of SCD patients in intensive care unit. However, its pathophysiology has long been poorly understood and therapeutic options are limited.

A major increase has been recently reported in the level of interleukin-6 (IL-6), unlike other main pro-inflammatory cytokines, in the sputum (or bronchoalveolar fluid) from SCD children during ACS, positively correlated with the severity of ACS. Also, the observations of a very rapidly favorable outcome after administration of tocilizumab (anti-human IL-6 receptor monoclonal antibody) in SCD patients hospitalized for ACS with or without SARS-CoV-2 infection, suggest that tocilizumab may be a key therapy for ACS.

ELIGIBILITY:
Inclusion Criteria:

1. SCD patient of all genotypes (SS, SC, S/β0 and S/β+)
2. Age ≥ 2 years old
3. Hospitalized for ACS, defined by the WHO as the association of fever and/or acute respiratory symptoms with a new pulmonary infiltrate on chest imaging, (X-ray, lung ultrasound, or CT scan)
4. Requiring supplemental oxygen ≥ 2 L/min for SpO2 ≥ 95% or non-invasive respiratory support (high flow nasal oxygen or continuous positive airway pressure or bilevel non-invasive ventilation) or invasive mechanical ventilation or ECMO, for less than 48 hours
5. Negative pregnancy test for girls or women of childbearing age
6. Freely given, informed and written consent of patient or legal representatives
7. Affiliation to the social security (or health insurance)
8. Effective contraception up to 3 months after the administration of treatment (tocilizumab or placebo)

Exclusion Criteria:

1. Impossibility to perform tocilizumab/placebo injection within the first 48 hours of supplemental oxygen and/or respiratory support (as defined in inclusion criteria n°4). If exchange transfusion is indicated at inclusion, it has to be performed before the injection of tocilizumab/placebo.
2. Known hypersensitivity to tocilizumab or its excipients
3. Known active current severe bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, and herpes zoster)
4. Immunization with a live/attenuated vaccine within the last 4 weeks
5. Immunomodulatory therapy, anti-rejection therapy, cell depleting therapies and investigational agents within the last 3 months
6. History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
7. History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower gastrointestinal disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower gastrointestinal conditions that might predispose a patient to perforations
8. Evidence of malignant disease or malignancies diagnosed within the last 3 years
9. Pregnancy or breastfeeding
10. Imminent and inevitable progression towards death in the opinion of the investigator
11. Absolute neutrophil count < 1.0 G/L or platelets < 50 G/L
12. ALT or AST > 5-fold the upper limit of normal
13. Glomerular Filtration rate (GFR) < 60 mL/min/1,73 m²
14. Current enrolment in another interventional research concerning a medicinal product for human use

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to successful weaning from both supplemental oxygen and any respiratory support | During hospitalization for ACS, from randomization until day 28 after randomization
  Successful weaning from both supplemental oxygen and any respiratory support, defined as SpO2 ≥ 95% without oxygen during the next 24 hours, and spontaneous breathing without any respiratory support (non-invasive or invasive) during the next 48 hours

SECONDARY OUTCOMES:
Adverse events during hospitalization and within 3 months following tocilizumab or placebo injection | Within 3 months after randomization
  Severe and not severe adverse events (including hypertension, hypersensitivity reactions, hypokalemia, neutropenia, thrombocytopenia, infections, pulmonary embolism/thrombosis, hepatic cytolysis, organ failure)
Time to discharge | From the date of randomization until the date of end of hospitalization, assessed up to 3 months
  Length of hospital stay
Mortality | Within 3 months after randomization
  Mortality
Need for transfusion | From the date of randomization until the date of end of hospitalization, assessed up to 3 months
  Need for red blood cell transfusion
Total number of red blood cell units received | From the date of randomization until the date of end of hospitalization, assessed up to 3 months
  Total number of red blood cell units received
Need for non-invasive ventilation (for patients without ventilatory support at inclusion) | From the date of randomization until the date of end of hospitalization, assessed up to 3 months
  Need for non-invasive ventilation (high flow nasal oxygen, continuous positive airway pressure, or bilevel non-invasive ventilation), for patients without ventilatory support at inclusion
Need for invasive ventilation (for patients without invasive ventilation at inclusion) | From the date of randomization until the date of end of hospitalization, assessed up to 3 months
  Need for invasive ventilation, for patients without invasive ventilation at inclusion
Readmission for vaso-occlusive crisis or ACS within 3 months following tocilizumab or placebo injection | Within 3 months after randomization
  Readmission for vaso-occlusive crisis or ACS within 3 months following tocilizumab or placebo injection
C-reactive protein (CRP), procalcitonin (PCT), plasma and sputum IL-6 levels 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  C-reactive protein (CRP), procalcitonin (PCT), plasma and sputum IL-6 levels 48 (+/- 12) hours after tocilizumab or placebo injection
Procalcitonin (PCT) level 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Procalcitonin (PCT) level 48 (+/- 12) hours after tocilizumab or placebo injection
Plasma IL-6 level 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Plasma IL-6 level 48 (+/- 12) hours after tocilizumab or placebo injection
Sputum IL-6 level 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Sputum IL-6 level 48 (+/- 12) hours after tocilizumab or placebo injection
Chest imaging improvement 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Improvement of chest imaging (chest X-ray or lung ultrasound) will be assessed by an investigator, who will have to choose between 3 possible answers: worsening, stability or improvement of ACS images.
Tocilizumab level in the plasma 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Tocilizumab level in the plasma 48 (+/- 12) hours after tocilizumab or placebo injection
Tocilizumab level in the sputum (or in the tracheal aspirations in case of invasive mechanical ventilation) 48 (+/- 12) hours after tocilizumab or placebo injection | 48 (+/- 12) hours after tocilizumab or placebo injection
  Tocilizumab level in the sputum (or in the tracheal aspirations in case of invasive mechanical ventilation) 48 (+/- 12) hours after tocilizumab or placebo injection

CONTACTS AND LOCATIONS:
Overall Officials: Slimane ALLALI, MD, PhD, Principal Investigator — Department of General Pediatrics and Sickle Cell Center, Necker-Enfants malades Hospital, Paris, France
Locations (1):
- Department of General Pediatrics and Sickle Cell Center, Necker-Enfants malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No